CLINICAL TRIAL: NCT05970055
Title: Prevalence and Associated Factors of Post-operative Nausea and Vomiting Among Adult Patients Undergoing Elective Surgery in DCSH, Dessie, Northeast Ethiopia, 2022
Brief Title: Prevalence and Associated Factors of Post-operative Nausea and Vomiting
Status: Completed | Type: Observational
Sponsor: Sara Timerga (Other)
Responsible Party: Sponsor-Investigator, Sara Timerga, Lecturer, Wollo University
Organization: Wollo University (Other)
Other Study IDs: WolloU
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PONV and Non PONV: PONV- patients who developed nausea and vomiting postoperatively Non PONV- patients who did not develop nausea and vomiting postoperatively
  Interventions: Procedure: elective surgery

INTERVENTIONS:
Procedure: elective surgery — All elective surgical procedures performed under the study period will be included.

SUMMARY:
Postoperative nausea and vomiting (PONV) is a surgical complication defined as any nausea, and vomiting with in the first 24-48 hours after surgery in inpatients. Nausea is an unpleasant feeling or desire to vomit without expulsive muscular movement, while vomiting is a forceful expulsion or reflux of the gastric contents through the mouth. Postoperative nausea and vomiting is one of the most common complication associated anesthesia and surgery. It is considered the most common cause of morbidity, and it has significant effects on patient satisfaction. In spite of recent development of anesthesia and surgical techniques, the incidence of PONV remains high. This common anesthetic and surgical side effect has been reported to increase patient dissatisfaction and can be just as distressing to patients as postoperative pain is.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting is caused by multiple factors; patient related, anesthesia and surgery related risk factors have been identified. Patient related factors include female gender post-puberty, nonsmoking status, history of PONV or motion sickness, and childhood after infancy and younger adulthood. Use of volatile anesthetics, nitrous oxide, large-dose neostigmine, or intraoperative or postoperative opioids are factors related to anesthesia, while the type of procedures like gynecologic, ophthalmological, ontological, thyroid surgery laparoscopic, abdominal surgery and duration of the procedure are some of surgery related risk factors.

The incidence of PONV for over multiple individual studies conducted around the world, has been estimated to be 25% to 30% and up to 80% in high risk groups. The incidence of PONV is estimated to range from 20%-36%.

Post-operative nausea and vomiting imposes multiple impacts on patients. The main one being a decrease satisfaction, but more importantly it leads to dehydration, electrolyte imbalance, aspiration of gastric secretions, esophageal rupture, bleeding, increased morbidity, and delayed discharge from hospital.

The study aimed to assess the incidence and associated factors of post-operative nausea and vomiting, which is believed to be a main contributing factor to dissatisfaction and delayed recovery seen in our country. The study was done from February to April 2022 in patients undergoing elective surgery at Dessie comprehensive specialized hospital, Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, who underwent elective surgery under anesthesia in the study period.

Exclusion Criteria:

* Patients who didn't gain their consciousness postoperatively, patients who underwent emergency surgery, patients who were re-operated on during the study period, surgical patients medical illness that predispose them to nausea and vomiting, and patients discharged before 24 hours postoperatively

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult, elective patients who underwent elective surgery under anesthesia at the Dessie comprehensive specialized hospital during the study period
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
post-operative nausea and vomiting | 24 hours
  Postoperative nausea and vomiting (PONV) is defined as any nausea, retching, or vomiting occurring during the first 24-48 h after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Timerga, Principal Investigator — Wollo University
Locations (1):
- Wollo Univeersity, Dessie, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD will depend on the requests.